CLINICAL TRIAL: NCT00246909
Title: Determination of the Minimal Clinically Important Difference (MCID) of the Patient Orientated Self Assessment Scale ReQuest TradeMark in Patients Suffering From Endoscopically Confirmed Gastroesophageal Reflux Disease (GERD), Grade A-D According to Los Angeles Classification Treated With Pantoprazole 40 mg o.d. or Placebo o.d. Over One Week.
Brief Title: Determination of the Minimal Clinically Important Difference After Treatment With Pantoprazole in Patients With Symptoms of Acid Reflux (Gastroesophageal Reflux Disease) (BY1023/M3-340)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Nycomed, Clinical Trial Operations
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY1023/M3-340
Record Dates: First submitted 2005-10-31; First posted 2005-11-01 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2011-06

CONDITIONS: Gastroesophageal Reflux
Keywords: Gastroesophageal Reflux; Gastroesophageal Reflux Disease; Pantoprazole
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Pantoprazole

INTERVENTIONS:
Drug: Pantoprazole

SUMMARY:
Gastroesophageal reflux disease (GERD) is a medical condition affecting the stomach and esophagus. GERD occurs when the lower esophageal sphincter does not close properly and stomach contents leaks back (refluxes) into the esophagus. GERD is one of the most common medical disorders, with estimates of up to 50% of adults reporting reflux symptoms daily. Proton pump inhibitors such as pantoprazole can relieve symptoms of GERD in a large proportion of patients.

Of particular interest in GERD is the assessment of symptom severity and quality of life, and the response of these parameters to treatment. Therefore, a questionnaire to assess GERD symptoms was developed (ReQuest TradeMark). An important point to consider when using such a questionnaire is to evaluate whether an observed difference in scores after a certain treatment represents a clinical effect.

The aim of this study is to determine the minimal clinically important difference (MCID) in patients diagnosed with GERD. During the study, the patients will complete a patient-orientated, self-assessed reflux questionnaire (ReQuest TradeMark). Endoscopy will be performed at the start of the study. The study duration consists of a baseline period (1 to 3 weeks) and a treatment period (8 weeks). During the first treatment week, the patients will receive either pantoprazole (tablet) or placebo once daily in the morning; for the following 7 treatment weeks all patients will receive pantoprazole. The study will provide further data on safety and tolerability of pantoprazole.

ELIGIBILITY:
Main inclusion criteria:

* In general good health other than gastroesophageal reflux disease (GERD)
* History of GERD-related symptoms for at least 6 months prior to inclusion into the study
* Endoscopically confirmed gastroesophageal reflux disease

Main exclusion criteria:

* Acute peptic ulcer and/or ulcer complications
* Systemic glucocorticoids or non-steroidal anti-inflammatory drugs (NSAIDs) including COX-2-inhibitors on more than 3 consecutive days within the previous 28 days; except regular intake of acetylsalicylic acid in dosages up to 163 mg/day
* Intake of Proton Pump Inhibitors and Histamine 2-receptor antagonists within the previous 14 days
* Intake of psychotropic medication, dyspepsia-inducing drugs, and anticholinergic agents
* Pregnant or nursing female patients; Non-pregnant, non-lactating female patients of childbearing potential who are not using reliable method of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2005-11; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
ReQuest(tm) scores after one week of treatment.

SECONDARY OUTCOMES:
other symptom assessments
safety.

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Heinze, PhD, Study Chair — Altana Pharma, D-78467 Konstanz, Germany
Locations (46):
- United States (46):
  - Altana Pharma/Nycomed, Alabaster, Alabama
  - Altana Pharma/Nycomed, Huntsville, Alabama
  - Altana Pharma/Nycomed, Mesa, Arizona
  - Altana Pharma/Nycomed, Tucson, Arizona
  - Altana Pharma/Nycomed, Little Rock, Arkansas
  - Altana Pharma/Nycomed, Anaheim, California
  - Altana Pharma/Nycomed, Los Angeles, California
  - Altana Pharma/Nycomed, Orange, California
  - Altana Pharma/Nycomed, Redwood City, California
  - Altana Pharma/Nycomed, San Diego, California
  - Altana Pharma/Nycomed, Wheat Ridge, Colorado
  - Altana Pharma/Nycomed, Torrington, Connecticut
  - Altana Pharma/Nycomed, Miami, Florida
  - Altana Pharma/Nycomed, Pembroke Pines, Florida
  - Altana Pharma/Nycomed, Hines, Illinois
  - Altana Pharma/Nycomed, Peoria, Illinois
  - Altana Pharma/Nycomed, Louisville, Kentucky
  - Altana Pharma/Nycomed, Baton Rouge, Louisiana
  - Altana Pharma/Nycomed, Shreveport, Louisiana
  - Altana Pharma/Nycomed, Bethesda, Maryland
  - Altana Pharma/Nycomed, Hollywood, Maryland
  - Altana Pharma/Nycomed, Laurel, Maryland
  - Altana Pharma/Nycomed, Reisterstown, Maryland
  - Altana Pharma/Nycomed, Towson, Maryland
  - Altana Pharma/Nycomed, Milford, Massachusetts
  - Altana Pharma/Nycomed, Jackson, Mississippi
  - Altana Pharma/Nycomed, Egg Harbor, New Jersey
  - Altana Pharma/Nycomed, Great Neck, New York
  - Altana Pharma/Nycomed, Johnson City, New York
  - Altana Pharma/Nycomed, Rochester, New York
  - Altana Pharma/Nycomed, Raleigh, North Carolina
  - Altana Pharma/Nycomed, Winston-Salem, North Carolina
  - Altana Pharma/Nycomed, Cincinnati, Ohio
  - Altana Pharma/Nycomed, Medford, Oregon
  - Altana Pharma/Nycomed, Duncansville, Pennsylvania
  - Altana Pharma/Nycomed, Philadelphia, Pennsylvania
  - Altana Pharma/Nycomed, Pittsburgh, Pennsylvania
  - Altana Pharma/Nycomed, Charleston, South Carolina
  - Altana Pharma/Nycomed, Chattanooga, Tennessee
  - Altana Pharma/Nycomed, Nashville, Tennessee
  - Altana Pharma/Nycomed, Houston, Texas
  - Altana Pharma/Nycomed, Salt Lake Citey, Utah
  - Altana Pharma/Nycomed, South Ogden, Utah
  - Altana Pharma/Nycomed, Fairfax, Virginia
  - Altana Pharma/Nycomed, Bellevue, Washington
  - Altana Pharma/Nycomed, Milwaukee, Wisconsin